CLINICAL TRIAL: NCT02429960
Title: Investigation of the Clinical Use of Different Analgesia-Monitors for Tracing Unconscious Pain Sensations During General Anesthesia
Brief Title: Comparison of Different Analgesia-Monitors in Tracing Unconscious Pain Sensations
Acronym: AMUPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Dr. med. Rainer Nitzschke, MD, Universitätsklinikum Hamburg-Eppendorf
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AMUPS-012013
Record Dates: First submitted 2015-04-08; First posted 2015-04-29 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Anesthesia
Keywords: Nociception; Analgesia; Intraoperative; Monitoring
MeSH Terms: conditions — Agnosia | interventions — Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Analgesia monitoring (Other): Remifentanil is increased step-by-step according to the study protocol. After ensuring a steady-state period of remifentanil infusion of at least 5 minutes, the standardized painful stimuli consisting of the intracutaneous pain model and tetanic stimulation for the time period of 30 s with 80 milliampere, 50 Hz are applied. All stimulations are accompanied by the measurement of the analgesic monitoring-devices (PhysioDoloris®, SPI® and AlgiScan®). Moreover the investigators measure and inspect changes in heart rate and blood pressure as well as occurrence of defensive movements of the patients.
  Interventions: Device: Analgesia monitor (PhysioDoloris®); Device: Analgesia monitor (SPI®); Device: Analgesia monitor (AlgiScan®); Drug: Remifentanil

INTERVENTIONS:
Device: Analgesia monitor (PhysioDoloris®) — Comparison of three different analgesia monitoring systems (PhysioDoloris®, SPI® and AlgiScan®).
Device: Analgesia monitor (SPI®) — Comparison of three different analgesia monitoring systems (PhysioDoloris®, SPI® and AlgiScan®).
Device: Analgesia monitor (AlgiScan®) — Comparison of three different analgesia monitoring systems (PhysioDoloris®, SPI® and AlgiScan®).
Drug: Remifentanil — Remifentanil will be increased step-by-step from 0.05 mcg/kg/min to 0.2 mcg/kg/min. After ensuring a steady-state period of remifentanil infusion of at least 5 minutes, the standardized painful stimuli will be applied.

SUMMARY:
Until today there is no standard-monitoring to specifically reflect the analgesic component of general anesthesia. Quality and safety of general anesthesia are of major clinical importance and can be improved by limiting the administration of opioid analgesics to the minimum dose needed. This study therefore examines the quality of three different monitoring techniques (PhysioDoloris, MetroDoloris, Lille, France, SPI (Surgical Plethysmographic Index), GE Healthcare, Helsinki, Finland and AlgiScan, IDMed, Marseille, France) in assessing the level of analgesia during general anesthesia. Therefore a standardized painful stimulus is applied under different levels of analgesic drugs. The monitor's indices are compared to clinical signs such as an increase in heart rate and blood pressure.

DETAILED DESCRIPTION:
This study aims to investigate the capability of different analgesia-monitors (PhysioDoloris, MetroDoloris, Lille, France, SPI (Surgical Plethysmographic Index), GE Healthcare, Helsinki, Finland and AlgiScan, IDMed, Marseille, France) in tracing unconscious pain sensations during general anesthesia. Many surgical procedures require general anesthesia. In order to induce hypnosis and analgesia, which are the main components of general anesthesia, the anesthetist usually combines a hypnotic drug with an opioid analgesic.

Until today, however, there is no standard-monitoring to specifically reflect the analgesic component of general anesthesia. Because over dosage as well as under dosage of opioids (e.g. remifentanil) may increase postoperative pain, the development of a depth-of-analgesia monitor is not only desirable but necessary. Quality and safety of general anesthesia are of major clinical importance and can be improved by limiting the administration of opioid analgesics to the minimum dose needed. This study therefore examines the quality of the monitoring technique, i.e. the sensitivity and specificity in assessing the level of analgesia during general anesthesia under standardized conditions.

Levels of analgesia are traditionally evaluated by clinical signs such as an increase in heart rate, blood pressure, lacrimation, sweating and defensive movements. Recent research has been able to demonstrate the possibility of assessment of the level of nociception-antinociception balance by applying a tetanic stimulation (30 s, 60 milliampere, 50 Hz) above the ulnar side of the wrist using a standard muscle relaxometer on the patients arm. In these investigations the stimulation led to a decrease of the vagal tonus resulting in changes in sinus arrhythmia and in a smaller area under the plethysmographic curve. Different devices were able to reflect a painful stimulus during propofol-remifentanil anesthesia. However, to the best of our knowledge, there are no data on the ability of the monitor-devices to detect a reproducible quantified painful stimulus under standardized conditions.

Bromm et al. thus established the intracutaneous pain model in the Department of Neurophysiology at the University-Hospital Hamburg-Eppendorf more than 20 years ago. This model involves removing a small core of epidermis from the skin on the pulp of the finger and placing an electrode directly in the vicinity of Aδ- and C-fiber terminals. Corresponding stimulation evokes clear pinprick pain of the patients. Utilizing Bromm et al.'s methodology, we actively contribute to the ongoing debate on the clinical use of analgesia-monitors in tracing unconscious sensation of pain during general anesthesia. For better comparability to previous studies the Bromm et al's methodology will be complemented by a measurement after a tetanic stimulation on each analgesic level.

The hypotheses will be examined in a prospective clinical study by means of tetanic stimulation, tested on presumably 30 elective patients. The study was approved by the Ethics committee of the Medical Board of the City of Hamburg, Germany and informed consent will be obtained from all patients. After induction of deep propofol sedation a laryngeal mask is inserted and sedation is maintained by continuous bispectral index-guided propofol-infusion. Next, remifentanil is increased step-by-step according to the study protocol.

After ensuring a steady-state period of remifentanil infusion of at least 5 minutes, the standardized painful stimuli consisting of the intracutaneous pain model and tetanic stimulation for the time period of 30 s with 80 milliampere, 50 Hz are applied. All stimulations are accompanied by the measurement of the analgesic monitoring-indices. Moreover the investigators measure and inspect changes in heart rate and blood pressure as well as occurrence of defensive movements of the patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Status I and II
* > 18 years
* Elective surgery in Urology/Ear Nose Throat under general anesthesia without the use of muscle relaxants

Exclusion Criteria:

* Diseases with impairment of sensitivity (diabetes, gout, polyneuropathy, peripheral arterial obstructive disease)
* Beta blocker and digitalis therapy
* Chronic pain therapy
* Pacemaker therapy
* Dermal diseases with affection of the forearm/hand

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the Pearson correlation coefficient between the dose of analgesic medication (remifentanil) on the one hand and the changes in heart rate, blood pressure and output of the analgesia monitoring systems on the other hand. | Observation for approximately 30 minutes after anesthesia induction

SECONDARY OUTCOMES:
Differences of sensitivity and specificity of the analgesia monitors in detecting a painful stimulus under different doses of remifentanil. | Observation for approximately 30 minutes after anesthesia induction
  Sensitivity and specificity of the analgesia monitors are compared to the sensitivity and specificity of the changes in heart rate and blood pressure after a painful stimulus.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Zoellner, Professor, Study Director — Department of Anesthesiology; Center of Anesthesiology and Intensive Care Medicine, Hamburg Eppendorf University Medical Center
Locations (1):
- Department of Anesthesiology; Center of Anesthesiology and Intensive Care Medicine, Hamburg Eppendorf University Medical Center, Hamburg, Germany

REFERENCES:
- See also: Publication of study results - Validation of Innovative Techniques for Monitoring Nociception during General Anesthesia — https://anesthesiology.pubs.asahq.org/article.aspx?articleid=2627427